CLINICAL TRIAL: NCT00040664
Title: A 48 Week, Phase II, Open-Label Multi-Cohort, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GW433908/Ritonavir QD and GW433908/Ritonavir BID When Administered to HIV-1 Infected, Antiretroviral Naive and Experienced, Pediatric Subjects 2-18 Years Old
Brief Title: A Clinical Study Of An Investigational Regimen Including Marketed HIV Drugs In HIV-1 Pediatric Subjects Ages 2-18 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APV 20003
Record Dates: First submitted 2002-07-05; First posted 2002-07-10 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: HIV Infection
Keywords: pediatrics; HIV; protease inhibitors; ritonavir; fosamprenavir; LEXIVA; AGENERASE; amprenavir
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; fosamprenavir

ARMS (3):
- 2 to 5 years (FPV/RTV) (Experimental): Two to five years. Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD)
  Interventions: Drug: ritonavir; Drug: fosamprenavir
- 6 to 11 years (FPV/RTV) (Experimental): Six to twelve years. Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD)
  Interventions: Drug: ritonavir; Drug: fosamprenavir
- 12 to 18 years (FPV/RTV) (Experimental): Twelve to Eighteen years. Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD)
  Interventions: Drug: ritonavir; Drug: fosamprenavir

INTERVENTIONS:
Drug: ritonavir — ritonavir oral capsules or oral solution
  Other Names: fosamprenavir
Drug: fosamprenavir — fosamprenavir oral suspension or tablet

SUMMARY:
This is a 48-week study to collect additional information on the safety, tolerability, pharmacokinetics, and antiviral activity of an investigational regimen (course of therapy) including FDA approved HIV drugs in HIV-infected patients 2 - 18 years old.

DETAILED DESCRIPTION:
A 48 Week, Phase II, Open-label, Multi-Cohort, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of GW433908/Ritonavir QD and GW433908/Ritonavir BID when Administered to HIV-1 Infected, Antiretroviral Naive and Experience Pediatric Subjects 2 to 18 Years Old

ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
* Inclusion Criteria:
* Male or females 2 to 18 years of age
* A female is eligible to enter and participate in this study if she is of:
* a. non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is pre-menarchial); or,
* b. child-bearing potential with a negative serum pregnancy test at screen, a negative urine pregnancy test on Day 1 and who agrees to use one of the following methods of contraception (any contraception method must be used consistently and correctly, i.e., in accordance with both the product label and the instructions of a physician). Note: hormonal contraceptives are not considered a sufficient form of contraceptive for this study.
* Complete abstinence from intercourse from 2 weeks prior to administration of study drugs, throughout the study and for 2 weeks after discontinuation of all study medications. Should a female subject of childbearing potential decide to become sexually active during the course of the study, she must be counselled and be willing to use one of the methods listed below:
* Double barrier contraception (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Any intrauterine device (IUD) with published data showing that the expected failure rate is less than 1% per year (not all IUDs meet this criterion)
* Any other method with published data showing that the lowest expected failure rate for that method is less than 1% per year. All subjects participating in this study should be counselled on the practice of safe/safer sex.
* Parent or legal guardian (and subject whenever possible) has the ability to understand and provide written informed consent for the subject to participate in the trial. Verbal witnessed assent must be obtained from the subject whenever possible.
* Screening plasma HIV-1 RNA > or =400copies/mL.
* Subject's who, in the investigator's opinion, and following resistance testing where appropriate, are able to construct an active NRTI backbone regimen consisting of 2 NRTIs.
* Subjects must meet one of the following criteria:
* ART-naïve subjects are defined as having had < 4 weeks (28 days) therapy with an NRTI, no previous therapy with an NNRTI and < 1 week therapy with an HIV PI.
* ART-experienced subjects are defined as having had greater than 4 weeks (28 days) therapy with any NRTI(s) and any length of therapy with any NNRTI(s) and/or a PI. PI-experienced subjects will be eligible if they have previously been treated with < three PIs, excluding AGENERASE. Prior therapy with a RTV boosted PI regimen will be considered as only 1 prior PI as long as the RTV dose was below that recommended for use of RTV as an antiretroviral agent. This specific criterion is not applicable to subjects in screening and/or enrolling after approval of Amendment No. 4. - For subjects screening and/or enrolling after the approval of Amendment No.4, PI naive subjects are defined as ART experienced subjects having less than one week of therapy with a PI and no prior experience with AGENERASE. Prior treatment with NNRTIs and NRTIs is permitted (however, subjects will NOT be permitted to receive concurrent NNRTI therapy while participating in this study)
* Exclusion Criteria:
* Prior history of having received amprenavir.
* Use of non-nucleoside reverse transcriptase inhibitor (NNRTI) therapy within 14 days of study Day 1 or anticipated need for concurrent NNRTI therapy during the study period.
* Have had an AIDS defining illness (acute CDC Category C event) within 28 days of screening.
* Pregnant or lactating.
* Non-nucleoside reverse transcriptase inhibitor therapy within 14 days prior to study drug administration or anticipated need for concurrent NNRTI therapy during the study period.
* Subjects who, in the investigator's opinion, are not able to comply with the requirements of the study.
* An acute CDC Category C event (per 1993/1994 classification) and/or serious bacterial infection(s) within 28 days prior to study drug administration.
* Presence of a malabsorption syndrome or other gastrointestinal dysfunction which might interfere with drug absorption or render the subject unable to take oral medication.
* Presence of any serious medical condition (e.g., hemoglobinopathy, chronic anemia,diabetes, cardiac dysfunction and hepatitis) which, in the opinion of the investigator, might compromise the safety of the subject.
* Current grade 2 or higher serum lipase within 28 days prior to study drug administration and/or history of clinically relevant pancreatitis within the previous 6 months. - Grade 3 or 4 transaminase levels (ALT and/or AST) within 28 days prior to study drug administration and/or clinically relevant hepatitis within the previous 6 months.
* Treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days of study drug administration or an anticipated need for such treatment within the study period.
* Treatment with immunomodulating agents (e.g., systemic corticosteroids, interleukins, interferons) or any agent with known anti-HIV activity (e.g., hydroxyurea or foscarnet) within 28 days of study drug administration.
* Treatment with any of the following medications within 28 days prior to receiving study medication or the anticipated need during the study:
* Amiodarone, astemizole, bepridil, bupropion, cisapride, clorazepate, clozapine, diazepin, dihydroergotamine, encainide, ergonovine, ergotamine, estazolam, flecainide, flurazepam, lovastatin, meperidine, methylergonovine, midazolam, pimozide, piroxicam, propafenone, propoxyphene, quinidine, rifabutin, simvastatin, terfenadine, triazolam, zolpidem (these drugs have been excluded for safety reasons).
* Carbamazepine, dexamethasone, phenobarbital, phenytoin, primidone, rifampin, St Johns Wort (these drugs have been excluded because they have the potential to decrease plasma protease inhibitor concentrations) - Systemic chemotherapeutic agents
* Treatment with other investigational drugs/therapies (note: treatments available through a Treatment IND or other expanded-access mechanism will be evaluated on a case-by-case basis in consultation with the sponsor) within 28 days prior to study drug administration
* History of drug or other allergy which, in the opinion of the investigator, contraindicates participation in the trial or known hypersensitivity to any study medications (e.g., documented hypersensitivity to a nucleoside analogue).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2002-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (16):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Richmond, Virginia
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Italy (7):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
- GSK Investigational Site, Rotterdam, Netherlands
- Portugal (2):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
- GSK Investigational Site, Bucharest, Romania
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohorts were recruited in parallel. All Age Cohorts were given the same treatment.
Pre-assignment Details: The overall study population consisted of 69 participants presented as "Overall Fosamprenavir (FPV)/ritonavir (RTV)" in the Participant Flow section. Furthermore, the Overall FPV/RTV participants are stratified by age cohorts (Arms 2-4).
Groups:
- Overall Fosamprenavir (FPV)/Ritonavir(RTV): Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD)
- 2-5 Years FPV/RTV: Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD), 2-5 years
- 6-11 Years FPV/RTV: Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD), 6-11 years
- 12-18 Years FPV/RTV: Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD), 12-18 years
Period: Overall Study
Arm/Group | Overall Fosamprenavir (FPV)/Ritonavir(RTV) | 2-5 Years FPV/RTV | 6-11 Years FPV/RTV | 12-18 Years FPV/RTV
Started | 69 (All (69) enrolled on QD; 10 switched to twice daily. Participant flow not collected for this group.) | 17 | 17 | 35
Completed | 16 | 4 | 4 | 8
Not Completed | 53 | 13 | 13 | 27
Not completed — Adverse Event | 12 | 3 | 2 | 7
Not completed — Lack of Efficacy | 9 | 2 | 3 | 4
Not completed — Insufficient CD4 response | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 2 | 0 | 2
Not completed — Protocol Violation | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 0 | 3 | 4
Not completed — Pregnancy | 3 | 0 | 0 | 3
Not completed — Medication adherence/compliance problems | 8 | 2 | 1 | 5
Not completed — Poor taste | 2 | 0 | 2 | 0
Not completed — Pharmacokinetic target not achieved | 2 | 1 | 0 | 1
Not completed — Change of formulation | 2 | 2 | 0 | 0
Not completed — Non-viability of oral suspension | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- FPV/RTV: Fosamprenavir (FPV) 700 mg tablets or 50 mg/mL oral suspension/ritonavir (RTV) 100 mg capsules or 80 mg/mL oral solution once daily (QD)
Arm/Group | FPV/RTV
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 35
  Black | 24
  East and South East Asian | 1
  American Hispanic | 8
  African Heritage | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Discontinued Treatment Due to Adverse Events
Description: The number of participants who prematurely discontinued study drug due to adverse events was tabulated. Data are summarized by individual adverse event.
Time Frame: Baseline through end of study (at least Week 168)
Population: Safety Population: all participants with documented evidence of having received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | FPV/RTV
Number analyzed (Participants) | 69
Participants
  Any event | 12
  Nausea | 3
  Vomiting | 3
  Stomach discomfort | 1
  Hyperglycaemia | 1
  Hypertriglyceridaemia | 1
  Blood alkaline phosphatase increased | 1
  Hodgkin's disease | 1
  Haemoptysis | 1

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies Per mL at Weeks 12, 48, 96, and 168 (Time to Loss of Virologic Response [TLOVR] Analysis)
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies per milliliter (mL) at Weeks 12, 48, 96, and 196. The percentage of participants with HIV-1 RNA <400 copies/mL at Weeks 12, 48, 96, 168 was determined by the TLOVR algorithm with stratification by the six randomization strata. TLOVR analysis categorizes participants by treatment response. Responders were participants with confirmed viral load <400copies/mL on two consecutive visits.
Time Frame: Weeks 12, 48, 96, and 168
Population: The Intent-to-Treat Exposed (ITT [E]) Population consisted of all subjects with documented evidence of having received at least one dose of study drug. Results are stratified by previous protease inhibitor (PI) experience. Participants with previous PI experience may respond differently to FPV.
Measure: Number; unit: percentage of participants
Groups:
- PI-Naive: Participants with equal to or less than 1 week of treatment with a Protease Inhibitor (PI)
- PI-Experienced: Participants treated with equal to or less than 3 PIs (any length of time)
Arm/Group | PI-Naive | PI-Experienced
Number analyzed (Participants) | 32 | 37
percentage of participants
  Week 12 | 22 | 20
  Week 48 | 16 | 16
  Week 96 | 13 | 11
  Week 168 | 11 | 7

3. Secondary Outcome: Median Change From Baseline HIV-1 RNA Values at Weeks 12, 48, 96, and 168 Visits
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in copies/mL at Weeks 12, 24, 48, 96, and 168. Change from Baseline was defined as the HIV-1 RNA level at Weeks 12, 24, 48, 96, and 168 minus the HIV-1 RNA level at Baseline.
Time Frame: Baseline and Weeks 12, 48, 96, and 168
Population: ITT-E Population. Results are stratified by previous PI experience. Participants with previous PI experience may respond differently to FPV.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | PI-Naive | PI-Experienced
Number analyzed (Participants) | 32 | 37
log10 copies/mL
  Week 12 | -2.85 [-3.12 to -2.54] | -2.03 [-3.02 to -0.64]
  Week 48 | -2.65 [-3.31 to -1.44] | -1.65 [-2.76 to -1.02]
  Week 96 | -2.52 [-3.14 to -1.42] | -1.76 [-2.91 to -0.57]
  Week 168 | -2.88 [-3.49 to -2.15] | -2.39 [-3.13 to -0.94]

4. Secondary Outcome: Median Change From Baseline in CD4+ Values at Week 12, 48, 96, and 168 Visits
Description: A blood sample was drawn to determine the CD4+ cell count at Weeks 24, 48, 96, and 168. Change from Baseline was defined as the CD4+ cell count at Weeks 24, 48, 96, and 168 minus the CD4+ cell count at Baseline.
Time Frame: Baseline and Weeks 12, 48, 96, and 168
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Cells/mm3
Groups:
- PI-Naive: Participants with equal to or less than 1 week of treatment with a PI
Arm/Group | PI-Naive | PI-Experienced
Number analyzed (Participants) | 32 | 37
Cells/mm3
  Week 12 | 95 [10 to 150] | 40 [-30 to 110]
  Week 48 | 150 [75 to 280] | 120 [0 to 240]
  Week 96 | 160 [55 to 280] | 40 [-180 to 180]
  Week 168 | 180 [10 to 430] | 0 [-220 to 200]

5. Primary Outcome: Number of Participants With Any Drug-related Grade 2 to 4 Adverse Event
Description: The number of participants with drug-related adverse events coded as Grade 2 (mild), Grade 3 (severe), or Grade 4 (life-threatening).
Time Frame: Baseline through end of study (at least Week 168)
Population: Safety Population: all participants with documented evidence of having received at least one dose of study drug
Measure: Number; unit: Participants
Groups:
- FPV Tablet: Fosamprenavir 700 mg tablets/ritonavir 100 mg capsules once daily
- FPV Oral Suspension: Fosamprenavir 50 mg/mL oral suspension/ritonavir 80 mg/mL oral solution once daily
Arm/Group | FPV Tablet | FPV Oral Suspension
Number analyzed (Participants) | 24 | 45
Participants
  All Grade 2-4 events | 7 | 14
  Vomiting | 0 | 5
  Diarrhea | 2 | 1
  Nausea | 2 | 1
  Blood alkaline phosphatase increased | 1 | 1
  Blood triglycerides increased | 1 | 0
  Abdominal pain | 0 | 1
  Benign salivary gland neoplasm | 0 | 1
  Blood cholesterol increased | 1 | 0
  Eosinophil count increased | 0 | 1
  Hemoptysis | 0 | 1
  Hyperglycemia | 0 | 1
  Hypertrichosis | 0 | 1
  Lipodystrophy acquired | 1 | 0
  Lipohypertrophy | 0 | 1
  Rash | 0 | 1
  Somnolence | 1 | 0
  Stomach discomfort | 1 | 0

6. Primary Outcome: Number of Participants With Grade 3 or 4 Treatment-emergent Laboratory Abnormalities
Description: The number of participants with Grade 3 (severe) or Grade 4 (life-threatening) laboratory abnormalities while on study treatment.
Time Frame: Baseline through end of study (at least Week 168)
Population: Safety Population: all participants with documented evidence of having received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | FPV/RTV
Number analyzed (Participants) | 69
Participants
  All parameters | 6
  Alanine aminotransferase | 2
  Aspartate aminotransferase | 3
  Cholesterol | 0
  Hyperglycemia | 0
  Hypoglycemia | 0
  Serum lipase | 0
  Triglycerides | 1
  Leucopenia | 1
  Neutropenia | 12
  Thrombocytopenia | 2
  Anemia | 1

7. Primary Outcome: Geometric Mean of Steady State Plasma Amprenavir (APV) Parameter: AUC(0-tau)
Description: Geometric mean is a type of "average" that indicates the central tendency of a set of values and is calculated by multiplying all the numbers in a set, and then taking the nth root of the resulting product. AUC(0-tau)=area under the concentration curve from time 0 to tau.
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: The Pharmacokinetic (PK) Parameter Population included all participants who underwent plasma PK sampling and provided full PK profiles with evaluable plasma APV PK parameter data; thus, the sample sizes were limited. Results are stratified by age cohort and formulation since these factors can impact PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: hours*micrograms/milliliter
Groups:
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 2-5 years
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 6-11 years
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 12-18 years
- FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years: FPV/RTV 1400/200 mg once daily (tablet), 12-18 years
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
hours*micrograms/milliliter | 47.3 [34.2 to 65.4] | 47.6 [27.0 to 84.0] | 75.5 [23.4 to 244] | 71.8 [10.6 to 486]

8. Primary Outcome: Geometric Mean of Steady State Plasma APV Parameter: Cmax
Description: Geometric mean is a type of "average" that indicates the central tendency of a set of values and is calculated by multiplying all the numbers in a set, and then taking the nth root of the resulting product. Cmax= concentration maximum.
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: The PK Parameter Population included all participants who underwent plasma PK sampling and provided full PK profiles with evaluable plasma APV PK parameter data; thus, the sample sizes were limited. Results are stratified by age cohort and formulation since these factors can impact PK profiles.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms/milliliter
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
micrograms/milliliter | 4.97 [3.76 to 6.58] | 5.07 [2.50 to 10.3] | 6.88 [4.31 to 11.0] | 7.70 [2.70 to 21.9]

9. Secondary Outcome: Number of Participants With APV Resistance Associated HIV-1 RNA Genotypic Mutations and Phenotypic Resistance at Time of Virologic Failure Not Present at Baseline
Description: A blood sample was drawn for participants failing to respond to therapy, and the mutations present in the virus were identified. For each participant, the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New mutations that developed at the time of virologic failure were tabulated by drug class. Virologic failure is defined as HIV-1 RNA greater than or equal to 400 copies/mL.
Time Frame: Time of virologic failure
Population: Participants in the ITT-E Population who met the virologic failure definition. Results are stratified by previous PI experience. Participants with previous PI experience may respond differently to FPV.
Measure: Number; unit: Participants
Arm/Group | PI-Naive | PI-Experienced
Number analyzed (Participants) | 32 | 37
Participants | 2 | 2

10. Primary Outcome: Median Steady State Plasma APV Tmax
Description: tmax: time after administration of the drug when maximum concentration is reached
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
hours | 1.04 [0.95 to 4.02] | 1.12 [0.75 to 2.07] | 1.08 [0.92 to 2.00] | 3.78 [1.00 to 4.00]

11. Primary Outcome: Geometric Mean of Steady State Plasma APV Parameter: CL/F
Description: Geometric mean is a type of "average" that indicates the central tendency of a set of values and is calculated by multiplying all the numbers in a set, and then taking the nth root of the resulting product. CL/F=apparent plasma clearance.
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters/minute/kilogram
Groups:
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 2-5 years vs. Historical Adult Data
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 6-11 years vs. Historical Adult Data
- FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years: FPV/RTV 30/6 mg/kg once daily (suspension), 12-18 years vs. Historical Adult Data
- FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years: FPV/RTV 1400/200 mg once daily (tablet), 12-18 years vs. Historical Adult Data
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
milliliters/minute/kilogram | 10.5 [7.62 to 14.5] | 10.6 [6.09 to 18.5] | 6.57 [2.08 to 20.7] | 4.95 [0.745 to 32.9]

12. Primary Outcome: Geometric Mean of Steady State Plasma APV Parameter: CL/F
Description: as for outcome 11
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: milliliters/minute
Arm/Group | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 3
milliliters/minute | 278 [41.2 to 1882]

13. Primary Outcome: Geometric Mean of Steady State Plasma APV Parameter: t1/2
Description: Geometric mean is a type of "average" that indicates the central tendency of a set of values and is calculated by multiplying all the numbers in a set, and then taking the nth root of the resulting product. t1/2=elimination half-life. t1/2=elimination half-life.
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
hours | 17.5 [11.1 to 27.7] | 13.6 [9.02 to 20.4] | 15.0 [7.93 to 28.2] | 14.9 [4.78 to 46.4]

14. Primary Outcome: Least Squares Mean of Plasma APV Parameter: AUC0-tau
Description: A blood sample was drawn on Week 4 over 24 hours (at 0, 1, 2, 4, 8, 12, and 24 hours post dosing). Ratio of geometric least squares mean (90% CI) are presented. Ctau=trough concentration. PK Parameters for QD and BID are compared with Historical adult data. Least squares mean (LSM) are the group means after having controlled for a covariate (i.e., holding it constant at some typical value of the covariate, such as its mean value). LSM is calculated by taking the average of the means within a treatment.
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: hours*micrograms/milliliters
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
hours*micrograms/milliliters | 0.695 [0.578 to 0.835] | 0.699 [0.577 to 0.848] | 1.11 [0.800 to 1.54] | 1.06 [0.761 to 1.47]

15. Primary Outcome: Least Squares Mean of Plasma APV Parameter: Cmax
Description: as for outcome 14
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: micrograms/milliliters
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
micrograms/milliliters | 0.663 [0.555 to 0.791] | 0.676 [0.560 to 0.814] | 0.917 [0.667 to 1.26] | 1.03 [0.747 to 1.41]

16. Primary Outcome: Least Squares Mean of Plasma APV Parameter: Ctau
Description: as for outcome 14
Time Frame: 0, 1, 2, 4, 8, 12, and 24 hours post dosing at Week 4.
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 2-5 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 6-11 Years | FPV/RTV 30/6 mg/kg Once Daily (Suspension), 12-18 Years | FPV/RTV 1400/200 mg Once Daily (Tablet), 12-18 Years
Number analyzed (Participants) | 10 | 9 | 3 | 3
microgram per milliliter | 0.716 [0.548 to 0.936] | 0.837 [0.663 to 1.06] | 0.963 [0.696 to 1.33] | 0.706 [0.568 to 0.878]

ADVERSE EVENTS:
Arm/Group | FPV/RTV
Serious Adverse Events (participants affected / at risk) | 19
Other Adverse Events (participants affected / at risk) | 63
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | FPV/RTV
Drug hypersensitivity (Immune system disorders) | 3/69
Measles (Infections and infestations) | 2/69
Pyrexia (General disorders) | 2/69
Appendicitis (Infections and infestations) | 1/69
Gastroenteritis (Infections and infestations) | 1/69
Pneumonia (Infections and infestations) | 1/69
Pneumonia bacterial (Infections and infestations) | 1/69
Aggression (Psychiatric disorders) | 1/69
Anxiety (Psychiatric disorders) | 1/69
Bipolar disorder (Psychiatric disorders) | 1/69
Borderline personality disorder (Psychiatric disorders) | 1/69
Depression (Psychiatric disorders) | 1/69
Impulse control disorder (Psychiatric disorders) | 1/69
Anemia (Blood and lymphatic system disorders) | 1/69
Hepatitis (Hepatobiliary disorders) | 1/69
Eye penetration (Injury, poisoning and procedural complications) | 1/69
Blood alkaline phosphatase increased (Investigations) | 1/69
Hyperglycemia (Metabolism and nutrition disorders) | 1/69
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/69
Headache (Nervous system disorders) | 1/69
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | FPV/RTV
Vomiting (Gastrointestinal disorders) | 28/69
Diarrhoea (Gastrointestinal disorders) | 18/69
Nausea (Gastrointestinal disorders) | 16/69
Abdominal pain (Gastrointestinal disorders) | 7/69
Abdominal pain upper (Gastrointestinal disorders) | 4/69
Dental caries (Gastrointestinal disorders) | 4/69
Upper respiratory tract infection (Infections and infestations) | 17/69
Bronchitis (Infections and infestations) | 12/69
Nasopharyngitis (Infections and infestations) | 11/69
Otitis media (Infections and infestations) | 8/69
Influenza (Infections and infestations) | 6/69
Oral herpes (Infections and infestations) | 4/69
Pharyngitis (Infections and infestations) | 4/69
Pharyngitis streptococcal (Infections and infestations) | 4/69
Sinusitis (Infections and infestations) | 4/69
Cough (Respiratory, thoracic and mediastinal disorders) | 16/69
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6/69
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5/69
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5/69
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4/69
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4/69
Rash (Skin and subcutaneous tissue disorders) | 10/69
Acne (Skin and subcutaneous tissue disorders) | 4/69
Pyrexia (General disorders) | 10/69
Headache (Nervous system disorders) | 17/69
Arthropod bite (Injury, poisoning and procedural complications) | 4/69
Lymphadenopathy (Blood and lymphatic system disorders) | 4/69
Conjunctivitis (Eye disorders) | 4/69
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.